CLINICAL TRIAL: NCT03478397
Title: Mixed-Methods Approach to Evaluate a mHealth Intervention to Increase Adherence to Triage of HPV+ Women Who Have Performed Self-collection
Brief Title: Evaluation of a mHealth Intervention to Increase Adherence to Triage of Self-collected HPV+ Women (ATICA Project)
Acronym: ATICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Estudio de Estado y Sociedad (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Deakin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-911
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-11

CONDITIONS: Patient Adherence
Keywords: cervical cancer prevention; self-collection HPV test; mHealth; Argentina
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent mHealth Intervention (Active Comparator): Women with HPV self-collected tests will receive a multicomponent intervention which includes SMS text messages to remind them to attend triage. In addition, CHWs will receive reminders via e-mails to contact women if after 60 days from the HPV-results HPV+ they have not performed triage.
  Interventions: Other: Multicomponent mHealth Intervention
- Usual Care (No Intervention): Women with HPV self-collected tests receive usual care. Upon opting for the HPV self-collected test, women will be instructed to go to the health care center in 30 days to pick up the results.

INTERVENTIONS:
Other: Multicomponent mHealth Intervention — Women with HPV self-collected tests will receive a multicomponent intervention which includes SMS text messages to remind them to attend triage. In addition, CHWs will receive reminders via e-mails to contact women if after 60 days from the HPV-results HPV+ they have not performed triage
  Arms: Multicomponent mHealth Intervention

SUMMARY:
Background: Cervical cancer is one of the leading causes of cancer death among women worldwide, with more than 85% of cases occurring in low- and middle-income countries. Human papillomavirus (HPV) screening allows for self-collection with the potential to increase coverage, but still requires triage to identify which HPV+ women need diagnostic and treatment procedures. However, achieving high levels of triage adherence can be challenging, especially among socially vulnerable women. The ATICA protocol (Application of Communication and Information Technologies to Self-Collection, for its initials in Spanish), aimed at evaluating the implementation strategy and the effectiveness of a multi-component mobile health (mHealth) intervention to increase adherence to triage among women with HPV+ self-collected tests. Methods: Researchers will use an effectiveness-implementation hybrid type I trial with a mixed-methods evaluation approach. A cluster randomized trial design including 200 community health workers (CHWs) will evaluate whether the mHealth intervention increases adherence to triage among HPV+ women who self-collected at home during a CHW visit within 120 days after a positive result. The intervention includes an initial mobile phone text message (SMS) alert and subsequent reminders sent to HPV+ women. For those who do not adhere to triage within 60 days of a positive HPV test, an email and SMS will be sent to the CHWs to promote contact with these women during home visits. Reserchers will use the Consolidated Framework for Implementation Research (CFIR) as an organizing and analytic framework to evaluate the implementation of the intervention while also drawing on Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM). Researchers will conduct a self-administered, semi-structured survey of CHWs, semi-structured interviews with local health authorities, and a survey of HPV+ women.

DETAILED DESCRIPTION:
Cervical cancer is a disease of health and gender inequalities, and is primarily a cancer of poor, socially vulnerable women. Even though it is almost entirely preventable, in Latin America it is the leading cause of cancer death among women.1 In Argentina, it is the second cause of female cancer death: every year 5,000 women are diagnosed with cervical cancer and more than 1,800 die from the disease.1 In this country, and generally across Latin America, high mortality is related to problems in the continuity of the prevention process, including low screening coverage and loss to follow-up, diagnosis, and treatment.2,3 New screening tests detect the presence of high-risk types of HPV which cause cervical cancer. HPV tests have important advantages over the Pap as a primary screening test, including higher sensitivity (over 90%)4 and a high negative predictive value,5 which allow reduced screening frequencies. Very importantly, through self-collection strategies, HPV testing can reduce barriers to screening and increase coverage.6 HPV self-collection is highly accurate,7 and is acceptable among women in different countries.8-11 However, HPV screening identifies women who are HPV+ (around 10%). Triage tests for HPV+ women determine those who need additional diagnostic procedures. While several triage methods are available for detecting precancerous lesions, including cytology and colposcopy,12 to date most such triage methods require HPV+ women to attend health centers to determine appropriate follow-up. Although adherence to follow-up and treatment is a widespread problem for cervical cancer programs in Latin America,2 evidence for interventions to improve adherence to follow-up is lacking.

The introduction of self-administered HPV testing in Jujuy has been successful in increasing primary cervical cancer screening coverage. Yet the proportion of self-collected HPV+ cases who currently undertake cytological triage within 120 days of screening is low (about 30%), which hinders the impact of the increased HPV screening coverage attained.

Aims of the study

1. To evaluate the effectiveness of a mHealth intervention targeted to women and health providers to increase adherence to cytological triage among self-tested HPV+ women compared to usual practice.
2. To identify and understand the processes and factors which contribute to the success of the mHealth intervention strategy (or lack thereof).

Setting Jujuy province is located in northwest Argentina and 85% of its population live in urban areas.19 The primary health care (PHC) system has 270 health centres and employs about 700 full-time CHWs who visit approximately 110,000 households twice a year for health-related tasks.

Since 2012, HPV-testing has been the primary CC screening test, available for women aged 30 years or older attending public health centres. Women are screened with HPV-testing every five years. Since 2014, HPV self-collection is offered during the CHW routine home visits. Women self-collect samples with a cervical sampler kit (Qiagen, Gaithersburg, MD, USA), which is comprised of a cervical brush, specimen container, and transport medium. Community health workers transport specimens at room temperature to health centres; from where they are sent to the provincial HPV laboratory to be analysed for 13 high-risk HPV types using hybrid-capture 2, following the manufacturer's instructions. According to the national guidelines,21 HPV-positive women with self-collected tests must go through cytology (triage Pap), and those HPV-positive women whose triage Paps are classified as atypical squamous cells of undetermined significance or worse (ASCUS+) are referred to colposcopy, then to biopsy if colposcopy images are classified as abnormal following the International Federation of Cervical Pathology and Colposcopy (IFCPC) classification.22 Women with histologically confirmed cervical intraepithelial neoplasia (CIN) of grade 2 or worse are referred to treatment.

All HPV-testing/diagnoses/treatments of women screened in the public health system are registered on the national screening information system (SITAM, for its initials in Spanish). Results of HPV tests and triage Paps are instantly available online to providers at public health establishments.

Setting The research will take place in the province of Jujuy, located in Northwest Argentina. Eighty-five percent of Jujuy's population lives in urban areas and the rate of mobile phone penetration was 82% of urban households in 201113 Jujuy has a high cervical cancer mortality rate (10.6 per 100.000 women during 2012-2014).

The Jujuy public health system includes a main hospital and 300 primary health care centers. For the uninsured, health services are provided free of cost. The Primary Health Care System (PHC) integrates approximately 700 paid full-time community health workers (CHWs) who twice yearly visit approximately 110,000 households for health-related tasks such as immunization and promoting maternal and child health.

Study design The study design follows the structure of an effectiveness-implementation hybrid type I trial14 and uses a mix-methods approach.

It combines a cluster randomized trial to evaluate the effectiveness of a multi-component mHealth intervention with a mixed methods approach involving quantitative and qualitative evaluations of the implementation using the RE-AIM15 and Consolidated Framework for Implementation Research (CFIR)16 frameworks.

The study will integrate quantitative and qualitative methods and follow Greene's typology of mixed-methods for convergence and complementarity.17 A formative research will be carried out to develop the framing and content of SMS messages (qualitative secondary method).

Then a pragmatic cluster randomized trial will be carried out to measure the effectiveness of the multi-component mHealth intervention in improving triage adherence among HPV+ women (quantitative primary method for Specific Aim 1).

Finally, during the post-intervention phase (Implementation evaluation for Specific Aim 2), a quantitative survey will be carried out to measure acceptability of the strategy by CHWs (quantitative secondary method), and semi-structured interviews (qualitative secondary methods) will be conducted among health authorities and health professionals,18 to receive feedback on their own perspectives and opinions about the intervention.19 HPV+ women will also be interviewed via a structured questionnaire (quantitative secondary method) to collect information about acceptability of the intervention, reasons for triage adherence/non-adherence, and their views about the strategy.

Formative research. Focus group discussions (FGD) will be carried out to explore women's opinions about how to frame and phrase SMS messages. Barriers women face in accessing triage will be explored, and the resulting information will be used to develop strategies CHWs can use to address them during the intervention. Drawing from FGD results, SMS messages will be designed and pilot tested with a validation protocol that has already been used in Argentina.20 Development of Automated Messaging system: an Automated System (AS) will be developed, which will then send SMS messages and e-mails based on data from the national Screening Information System (SITAM). This AS will will work in an asynchronous manner. In order to avoid sending a SMS message to the wrong person, an identity verification process will be initiated. Only matching data will be classified as "valid" and receive subsequent SMS messages. E-mails sent to CHWs will not include personal information about women, but a secure link to registries of women to be viewed in SITAM. SMS messages and e-mails will comply with security procedures.

Intervention: cluster-randomized trial. Approximately 200 CHWs from Jujuy's PHC will be randomized into two groups: 1) mHealth Intervention (MH) Group: Women with positive self-collected tests will receive a multi-component intervention. HPV+ women will receive periodic SMS messages during the first month after registration of self-collection test result in SITAM, notifying them that test results are available and they should go to the health center. In addition, CHWs will receive an e-mail and SMS message prompting them to visit those HPV+ women who, at 60 days since availability of the HPV result in SITAM, have not attended triage. CHWs will be asked to confirm receipt of the e-mail for monitoring project processes. Within 15 days of being notified, CHWs will visit these HPV+ women, for an in-person reminder and counseling about the importance of attending health centers and have triage performed. 2) Usual Care (UC) Group: Women with positive self-collected tests will receive usual care, i.e., women opting for self-collection will be instructed to go the health center in 30 days to pick up results.

Hypothesis: Adherence to triage will be higher in the MH intervention group compared to women receiving UC.

Study procedures. CHWs from both groups will identify eligible women and invite them to participate in the study during their routine home visits. Once women have performed HPV-self collection, CHWs will screen for eligibility criteria, including use of mobile phones. Those women who use a mobile phone will be explained the study objectives and will be invited to participate in the study. Women accepting to participate will be asked to provide a telephone number. Based on previous studies,21,22 the investigators expect approximately 85% of women will provide a telephone number; with 70% providing their own personal mobile phone.

MH Group: CHWs will carefully explain participants the sequence of SMS messages to be received depending on the Test results, and how they should proceed after reception of the SMS messages. If the woman does not have a personal phone, she will be asked if she is willing to be contacted and receive the proposed SMS messages on a shared phone. CHWs will inform women about the nature and content of the SMS messages to be received. They will also explain that if they have not performed triage 60 days after a positive test results they will come back for an in-person visit. Therefore, consent to participate also means women agreement to be contacted and to receiving SMS messages, even if phones are shared by several family members.

Upon SITAM registration of the HPV result, a first SMS message will be sent requiring women a confirmatory reply with their id number. This confirmatory approach to assure a patient's identity has been used and proved effective in other studies.22,23 After confirmation, women will receive a second SMS message with different information depending on their HPV status: if HPV-, they will be informed about the result and date of next screening; if HPV+, they will be informed that test results are available at the health center. Women will know in advance that this SMS message will mean they are HPV+. During the first four weeks after registration of a HPV result in SITAM, a SMS message will be sent weekly unless a Pap result is registered in SITAM. Sixty days after the date of registration of the HPV test result in SITAM, CHWs will receive an e-mail and SMS message informing them that there are HPV+ women who have not had Pap triage (if this is the case). The e-mail will contain a secure link to the list of HPV+ women to be visited. CHWs will be asked to confirm receipt of the e-mail for monitoring project processes. CHWs will visit these HPV+ women within 15 days of being notified, for an in-person reminder and counseling about the importance of attending health centers and have triage performed. CHW visit information will be recorded, including visit attempts, date of visit and issues addressed during counseling.

UC care group: Once women have agreed to participate in the project, CHWs will provide UC counseling using specific24 standard provincial protocol and materials. They will inform women that they should go to the health center in a month to get their test results.

Randomization and sample size: All CHWs (clusters) (approximately 700) of the Jujuy province offer self-collection and will be eligible to participate in the study. After classifying them into four groups according to gender and urban/rural setting, a stratified sample of 240 CHWs will be randomly selected with allocation proportional to strata. Selected CHWs will be invited to participate in the study following the order defined by the random list until 200 are enrolled. Enrolled CHWs will be randomly allocated to the MH or the UC group (3:2 ratio). Blinding of intervention and outcome assessments is not feasible due to the characteristics of the study. Primary outcome: The target sample size (120 CHWs in the MH group and 80 CHWs in the UC group, each one providing 2 HPV+ women) will have 97% power to detect a 20% triage difference between the two groups when the control group has a 30% triage in a 120-days period (two-sided test, alpha=0.05). Correlation induced by the CHWs was included in power calculations assuming an intra-class correlation coefficient of 0.10. Secondary outcome: Under the same assumptions, the proposed sample size will have 90% power to detect a difference of 10% in triage between groups when the control group has a 15% triage by day 60.

Analysis plan: All analysis will be conducted in an intention-to-treat basis, i.e. an enrolled woman with a positive HPV result will be considered in the study group assigned to her CHW, regardless of adherence of the CHW to the intervention or the number of SMS messages delivered to the woman. The effect of the multi-component mHealth intervention on the primary outcome will be assessed using a generalized estimating equations approach. The model, logit link, and binomial distribution will include trial group as fixed effect and CHWs as the clustering variable. Potential modification of the effect of the intervention due to rural/urban location of the woman and CHW gender will be evaluated, additionally including these factors and their interactions with study group in the former model. Baseline women factors will be compared between groups. Factors showing clear unbalance between arms will be included in the model proposed above to adjust for potential confounding. The same approach will be used to estimate the intervention effect on the secondary outcome. An interrupted time series approach will be used to explore the differential impact of each component of the intervention (SMS messages to women from day 1-59, SMS message and e-mail to CHWs by day 60) on the total number of women with triage at each week. Baseline for each woman will be defined as the day the HPV tests results are recorded in SITAM. Segmented regression will be used to assess the trend of the outcome in each period (1-59; 60-120 days) and any potential discontinuity (change in level or profile) in the time series of the intervention group compared to the control group. A linear model accounting for the autocorrelation of the data and including period (1-59; 60-120 days), intervention indicator (yes/no), and functions of time before and after the breakpoint (date when the second component starts) will be fitted. Given that the number of HPV+ women with triage is not expected to follow a linear trend with time, smooth functions (spline) of time will be used to model the relation between outcome and time in each study group. Under the assumption that the trend in the outcome would remain unchanged in the absence of the second component, this approach will allow investigators to describe the counterfactual curve expected in the intervention group had the second component not been implemented. Analyses will be conducted using STATA and/or SAS. The trial will follow the CONSORT extension for cluster randomized trials reporting guidelines 25.

ELIGIBILITY:
Inclusion Criteria:

In the Randomized Controlled Trial we will recruit a minimum of 4000 women, aged 30 and older living in the province of Jujuy, Argentina.

Inclusion criteria are:

1. Having performed self-collection of HPV-testing.
2. Mentally competent to understand the consent form.
3. Able to communicate with study staff.
4. Being able to provide a mobile phone telephone number.

Exclusion Criteria:

* Current pregnancy.
* Women with Mental disability.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5389 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvina Arrossi, Phd, Principal Investigator — CEDES/CONICET
Locations (1):
- Multiple facilities, San Salvador de Jujuy, Jujuy Province, Argentina

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Murillo R, Almonte M, Pereira A, Ferrer E, Gamboa OA, Jeronimo J, Lazcano-Ponce E. Cervical cancer screening programs in Latin America and the Caribbean. Vaccine. 2008 Aug 19;26 Suppl 11:L37-48. doi: 10.1016/j.vaccine.2008.06.013. PMID 18945401
- [Background] Arrossi S, Paolino M, Thouyaret L, Laudi R, Campanera A. Evaluation of scaling-up of HPV self-collection offered by community health workers at home visits to increase screening among socially vulnerable under-screened women in Jujuy Province, Argentina. Implement Sci. 2017 Feb 13;12(1):17. doi: 10.1186/s13012-017-0548-1. PMID 28193227
- [Background] Cuzick J, Arbyn M, Sankaranarayanan R, Tsu V, Ronco G, Mayrand MH, Dillner J, Meijer CJ. Overview of human papillomavirus-based and other novel options for cervical cancer screening in developed and developing countries. Vaccine. 2008 Aug 19;26 Suppl 10:K29-41. doi: 10.1016/j.vaccine.2008.06.019. PMID 18847555
- [Background] Dillner J, Rebolj M, Birembaut P, Petry KU, Szarewski A, Munk C, de Sanjose S, Naucler P, Lloveras B, Kjaer S, Cuzick J, van Ballegooijen M, Clavel C, Iftner T; Joint European Cohort Study. Long term predictive values of cytology and human papillomavirus testing in cervical cancer screening: joint European cohort study. BMJ. 2008 Oct 13;337:a1754. doi: 10.1136/bmj.a1754. PMID 18852164
- [Background] Gok M, Heideman DA, van Kemenade FJ, Berkhof J, Rozendaal L, Spruyt JW, Voorhorst F, Belien JA, Babovic M, Snijders PJ, Meijer CJ. HPV testing on self collected cervicovaginal lavage specimens as screening method for women who do not attend cervical screening: cohort study. BMJ. 2010 Mar 11;340:c1040. doi: 10.1136/bmj.c1040. PMID 20223872
- [Background] Arbyn M, Verdoodt F, Snijders PJ, Verhoef VM, Suonio E, Dillner L, Minozzi S, Bellisario C, Banzi R, Zhao FH, Hillemanns P, Anttila A. Accuracy of human papillomavirus testing on self-collected versus clinician-collected samples: a meta-analysis. Lancet Oncol. 2014 Feb;15(2):172-83. doi: 10.1016/S1470-2045(13)70570-9. Epub 2014 Jan 14. PMID 24433684
- [Background] Arrossi S, Thouyaret L, Herrero R, Campanera A, Magdaleno A, Cuberli M, Barletta P, Laudi R, Orellana L; EMA Study team. Effect of self-collection of HPV DNA offered by community health workers at home visits on uptake of screening for cervical cancer (the EMA study): a population-based cluster-randomised trial. Lancet Glob Health. 2015 Feb;3(2):e85-94. doi: 10.1016/S2214-109X(14)70354-7. PMID 25617202
- [Background] Giorgi Rossi P, Marsili LM, Camilloni L, Iossa A, Lattanzi A, Sani C, Di Pierro C, Grazzini G, Angeloni C, Capparucci P, Pellegrini A, Schiboni ML, Sperati A, Confortini M, Bellanova C, D'Addetta A, Mania E, Visioli CB, Sereno E, Carozzi F; Self-Sampling Study Working Group. The effect of self-sampled HPV testing on participation to cervical cancer screening in Italy: a randomised controlled trial (ISRCTN96071600). Br J Cancer. 2011 Jan 18;104(2):248-54. doi: 10.1038/sj.bjc.6606040. Epub 2010 Dec 21. PMID 21179038
- [Background] Leniz J, Barriga MI, Lagos M, Ibanez C, Puschel K, Ferreccio C. HPV vaginal self-sampling among women non-adherent to Papanicolaou screening in Chile. Salud Publica Mex. 2013 Apr;55(2):162-9. doi: 10.1590/s0036-36342013000200007. PMID 23546407
- [Background] Zehbe I, Moeller H, Severini A, Weaver B, Escott N, Bell C, Crawford S, Bannon D, Paavola N. Feasibility of self-sampling and human papillomavirus testing for cervical cancer screening in First Nation women from Northwest Ontario, Canada: a pilot study. BMJ Open. 2011 Feb 26;1(1):e000030. doi: 10.1136/bmjopen-2010-000030. PMID 22021733
- [Background] WHO Guidelines for Screening and Treatment of Precancerous Lesions for Cervical Cancer Prevention. Geneva: World Health Organization; 2013. Available from http://www.ncbi.nlm.nih.gov/books/NBK195239/ PMID 24716265
- [Background] Instituto Nacional de Estadísticas y Censos (INDEC). Encuesta Nacional sobre Acceso y Uso de Tecnologías de la Información y la Comunicación (ENTIC). Resultados del tercer trimestre de 2011. Buenos Aires: INDEC; 2012. Available from: http://www.indec.gov.ar/uploads/informesdeprensa/entic_06_13.pdf (accessed October 3, 2015).
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Sofaer S. Qualitative methods: what are they and why use them? Health Serv Res. 1999 Dec;34(5 Pt 2):1101-18. PMID 10591275
- [Background] Teddlie C, Tashakkori A. Major issues and controversies in the use of mixed methods in the social and behavioral sciences. In Tashakkori A & Teddlie C (Eds.). Handbook of mixed methods in the social and behavioral sciences (pp. 3-50). Thousand Oaks, CA: Sage; 2003
- [Background] Diez-Canseco F, Zavala-Loayza JA, Beratarrechea A, Kanter R, Ramirez-Zea M, Rubinstein A, Martinez H, Miranda JJ. Design and Multi-Country Validation of Text Messages for an mHealth Intervention for Primary Prevention of Progression to Hypertension in Latin America. JMIR Mhealth Uhealth. 2015 Feb 18;3(1):e19. doi: 10.2196/mhealth.3874. PMID 25693595
- [Background] Cormick G, Ciganda A, Cafferata ML, Ripple MJ, Sosa-Estani S, Buekens P, Belizan JM, Althabe F. Text message interventions for follow up of infants born to mothers positive for Chagas disease in Tucuman, Argentina: a feasibility study. BMC Res Notes. 2015 Sep 29;8:508. doi: 10.1186/s13104-015-1498-9. PMID 26419230
- [Background] Bobrow K, Brennan T, Springer D, Levitt NS, Rayner B, Namane M, Yu LM, Tarassenko L, Farmer A. Efficacy of a text messaging (SMS) based intervention for adults with hypertension: protocol for the StAR (SMS Text-message Adherence suppoRt trial) randomised controlled trial. BMC Public Health. 2014 Jan 11;14:28. doi: 10.1186/1471-2458-14-28. PMID 24410738
- [Background] Rubinstein A, Miranda JJ, Beratarrechea A, Diez-Canseco F, Kanter R, Gutierrez L, Bernabe-Ortiz A, Irazola V, Fernandez A, Letona P, Martinez H, Ramirez-Zea M; GISMAL group. Effectiveness of an mHealth intervention to improve the cardiometabolic profile of people with prehypertension in low-resource urban settings in Latin America: a randomised controlled trial. Lancet Diabetes Endocrinol. 2016 Jan;4(1):52-63. doi: 10.1016/S2213-8587(15)00381-2. Epub 2015 Dec 1. PMID 26653067
- [Background] Cuberli M, Arrossi S. Consejería para la prevención del cáncer de cuello de útero. Propuestas para una mejor comunicación con las mujeres durante el tamizaje, seguimiento y tratamiento. Buenos Aires: Instituto Nacional del Cáncer (INC); 2013.
- [Background] Campbell MK, Piaggio G, Elbourne DR, Altman DG; CONSORT Group. Consort 2010 statement: extension to cluster randomised trials. BMJ. 2012 Sep 4;345:e5661. doi: 10.1136/bmj.e5661. No abstract available. PMID 22951546
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] Arrossi S, Paolino M, Orellana L, Thouyaret L, Kohler RE, Viswanath K. Mixed-methods approach to evaluate an mHealth intervention to increase adherence to triage of human papillomavirus-positive women who have performed self-collection (the ATICA study): study protocol for a hybrid type I cluster randomized effectiveness-implementation trial. Trials. 2019 Feb 26;20(1):148. doi: 10.1186/s13063-019-3229-3. PMID 30808379

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Effectiveness trial women recruitment took place between December 4, 2018, and July 31, 2019.
  HPV self-collection is offered during the CHW routine home visits. During the visit, CHWs identified eligible women and invited them to participate.
Pre-assignment Details: All CHWs were assigned to the trial arms at the same time guaranteeing allocation concealment. Regarding women's consent, the CHWs were instructed to invite the woman and seek consent before disclosing their group allocation.
Period: Overall Study
Arm/Group | Multicomponent mHealth Intervention | Usual Care
Started (Eligible women invited) | 3272 | 2117
Women Accepted to Participate | 3241 | 2110
Completed | 3241 | 2110
Not Completed | 31 | 7
Not completed — Refused to participate | 31 | 7

BASELINE CHARACTERISTICS:
Population: HPV-positive women
Groups:
- Total: Total of all reporting groups
Arm/Group | Multicomponent mHealth Intervention | Usual Care | Total
Number analyzed (Participants) | 445 | 292 | 737
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 445 | 292 | 737
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 445 | 292 | 737
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Argentina | 445 | 292 | 737
Triage Pap smear [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Women With Triage Pap Smears at 120 Days After HPV Results
Description: The percentage of women with triage Pap smears at 120 days after HPV results are registered in the national screening information system (SITAM). This will allow measurement of the overall effect of the multi-component intervention including two periods: a) the 60 day period between the Test results and the SMS message and e-mail sent to Community Health Workers (CHW) (days 1-59); and b) the 60 day period between the SMS message and e-mail sent to CHWs and triage measurement (days 60-120)
Time Frame: 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | Multicomponent mHealth Intervention | Usual Care
Number analyzed (Participants) | 445 | 292
Participants | 314 | 163

2. Secondary Outcome: Percentage of Women With Triage Pap Smears at 60 Days After HPV Results
Description: The percentage of women with triage Pap smears at 60 days after HPV results are registered in SITAM (days 1-59). This outcome will allow us to measure the individual effect of the SMS messages sent to women (before CHWs receive prompts to contact non compliant HPV+ women).
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Multicomponent mHealth Intervention | Usual Care
Number analyzed (Participants) | 445 | 292
Participants | 242 | 101

ADVERSE EVENTS:
Time Frame: Through study completion, for 1 year.
Description: None untoward or unfavorable medical occurrences were detected related to the participant's participation in the research.
Arm/Group | Multicomponent mHealth Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/3272 | 0/2117
Serious Adverse Events (participants affected / at risk) | 0/3272 | 0/2117
Other Adverse Events (participants affected / at risk) | 0/3272 | 0/2117

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT03478397/Prot_SAP_000.pdf